CLINICAL TRIAL: NCT01148121
Title: Assessment of Bone Density and Bone Turnover Markers in Patients With Down Syndrome and Comparison to the Ts65Dn Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 113810
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Skeletal Status Assessment of a Down Syndrome Population — The investigators hypothesize that the bone deficits seen in Down Syndrome patients are similar to the phenotype seen in the down syndrome mouse model (Ts65Dn).The bone turnover markers, CBC, and DXA scan results will be used to assess the skeletal status of the down syndrome patients. This data will form the basis to establish the Ts65Dn as a reasonable proxy for pathogenesis and treatment in humans.

SUMMARY:
This study may provide information that may serve as the foundation for a larger research study to address issues regarding the causes, diagnosis, and treatment of osteoporosis in the Down syndrome patient population.

DETAILED DESCRIPTION:
Osteoporosis is responsible for more than 1.5 million fractures and $14 billion in medical care costs annually (U.S Dept of Health and Human Services data, 2006). Down syndrome is an independent risk factor for osteopenia/osteoporosis. Increases in life expectancy as well as costly morbidity following fracture are reasons for further investigation of osteoporosis and prevention in this population. Etiology for low bone density is presently unknown in this population but may be related to unique genes on chromosome 21 which alter the biochemistry of bone metabolism or change the gonadal, thyroid and parathyroid function to alter bone formation and/or resorption. There are no published data on the measurement of bone turnover markers in the Down syndrome population; therefore we will measure and accrue this information and compare to our Ts65Dn data, as described later in this protocol.

This pilot study will serve as the foundation for a larger translational research grant which will address multiple issues regarding the pathogenesis, diagnosis and treatment of osteoporosis in the Down syndrome patient population and the Down syndrome mouse model (Ts65Dn). The data has the potential to improve our fundamental understanding of osteoporosis pathogenesis and treatment in the Down syndrome patient with potential applications to treatment in the general population.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females of all races and ethnicities
* Age 18 or older and current clinical diagnosis of Down Syndrome

Exclusion Criteria:

* No legally authorized representative (if applicable) willing to provide informed consent. Any condition the investigator determines will put the subject at risk by participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Ts65DN pathogenesis proxy | 1 year
  The bone turnover markers, Complete Blood Count (CBC) and the Duel Energy X-ray (DXA) scan results will be used to assess the skeletal status of the Down syndrome patients. This data will form the basis to establish the Ts65Dn as a reasonable proxy for pathogenesis and treatment in humans.

CONTACTS AND LOCATIONS:
Overall Officials: Kent D McKelvey, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States